CLINICAL TRIAL: NCT04848688
Title: Efficacy and Safety of Moxidectin in Comparison to Ivermectin Against Strongyloides Stercoralis Infection in Adults: a Randomized Controlled Non-inferiority Trial
Brief Title: Efficacy and Safety of Moxidectin Versus Ivermectin Against Strongyloides Stercoralis
Acronym: StrongMoxi_KH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jennifer Keiser (Other)
Collaborators: National Centre for Parasitology, Entomology and Malaria Control, Cambodia (Other)
Responsible Party: Sponsor-Investigator, Jennifer Keiser, Prof. Jennifer Keiser, PhD, Swiss Tropical & Public Health Institute
Organization: Swiss Tropical & Public Health Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4
Record Dates: First submitted 2021-04-08; First posted 2021-04-19 (Actual); Results first posted 2024-01-24 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Strongyloides Stercoralis Infection
MeSH Terms: interventions — moxidectin; Ivermectin

STUDY DESIGN:
Intervention Model Description: Parallel study with 2 treatment arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded (Participant and Care provider) Additionally, the principal investigator and the statistician will be blinded.
  PK substudy is single-blinded (Participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moxidectin (Experimental): 8 mg Moxidectin at day 0 administered orally
  Interventions: Drug: Moxidectin 2 mg; Drug: Placebo
- Ivermectin (Experimental): 200 ug/kg Ivermectin at day 0 administered orally
  Interventions: Drug: Ivermectin 3 mg; Drug: Placebo

INTERVENTIONS:
Drug: Moxidectin 2 mg — Monotherapy, oral administration, single-dose, fixed-dose, 4 tablets of 2 mg each to yield an 8 mg final dose.
  Arms: Moxidectin
Drug: Ivermectin 3 mg — Monotherapy, oral administration, single-dose, weight dependent, The number of tablets will be adjusted according to the patients' weight to yield 200 ug/kg final dose.
  Arms: Ivermectin
Drug: Placebo — Monotherapy, oral administration, single dose, matching number of tablets to either moxidectin or ivermectin

SUMMARY:
The study is an extension to the study StrongMoxi NCT04056325 and entails modifications based on the outcome of NCT04056325 part A.

The study is a phase 3, double-blinded and randomized clinical trial conducted in Cambodia. It aims at providing evidence on efficacy, safety and pharmacokinetic measures of 8 mg of moxidectin compared to 200 μg/kg ivermectin in adults infected with S. stercoralis. The efficacy of the treatment will be assessed by collecting three stool samples once per-treatment and once 21-28 days post-treatment. The stool samples will be analyzed by a quantitative duplicate Baermann assay.

DETAILED DESCRIPTION:
The study is a phase 3 trial and will determine the efficacy and safety of:

8 mg of moxidectin in comparison to the standard treatment dose of ivermectin (200 μg/kg) in adults infected with S. stercoralis and to measure moxidectin disposition in adults using a microsampling device.

Our primary objective is to demonstrate non-inferiority in terms of cure rate (CR) against S. stercoralis in adults of an oral 8 mg of moxidectin compared to 200 μg/kg of ivermectin.

The secondary objectives of the trial are:

1. to evaluate the safety and tolerability of moxidectin
2. to compare the larval reduction rate (LRR) of the two different treatment groups against S. stercoralis
3. to evaluate the CRs of the different treatment drugs and regimens against soil-transmitted helminths (STH) co-infections.
4. to investigate potential extended effects on follow-up helminth prevalence at 42-49 and 63-70 days post-treatment
5. to relate socioeconomic characteristics (SES), access to sanitation, water facilities, hygiene to baseline infection intensity.
6. to determine the larval excretion pattern till day 70 in the moxidectin treatment arm, determined at every second day between day zero and 70 post-treatment in a subset of 50 adults.
7. to determine the origin of the remaining worm burden after treatment to treatment failure and reinfection based on genetic profiling.

Three stool samples will be collected at baseline analysed in duplicates by a quantitative Baermann method for S. stercoralis infection. Co-infection with other Helminths species will be identified using duplicate Kato-Katz thick smears on two stool samples. The medical history of the participants will be assessed with a standardized questionnaire, in addition to a clinical and physical examination carried out by the study physician shortly before the treatment day. Each participant will be asked to provide a finger-prick blood sample for haemoglobin measurements at baseline. Enrolled participants will be treated with either 8 mg of moxidectin or with the standard treatment ivermectin (200 μg/kg). The adults will be interviewed a) before treatment, 2-3 and 24 hours as well as 14-21, 42-49 and 63-70 days after treatment about the occurrence of adverse events. The efficacy of the treatment will be determined 14-21 days of post-treatment. All stool samples will be examined with quantitative sixtuplicate Baermann assays and quadruplet Kato-Katz thick smears. At 42-49 and 63-70 days post-treatment another three stool samples will be collected and quantified for S. stercoralis larvae using Baermann assay to assess potential long-term benefits of the study drugs and treatment regimen. Of 50 adults in the moxidectin arm only, additional stool samples will be collected every second day between treatment and 70 days post treatment to evaluate larval secretion patterns.

To all participating households, a brief questionnaire will be administered assessing information on socioeconomic characteristics (SES) and access to sanitation, water facilities, and hygiene behaviour.

An available case analysis (full analysis set according to the intention to treat principle) will be performed, including all participants with primary endpoint data.

CRs will be calculated as the percentage of larvae-positive subjects at baseline who become larvae-negative after treatment, assessed 14-21 days post-treatment by sextuplicate Baermann. Uncertainty estimates around the differences among CRs will be assessed using melded confidence intervals with mid-p correction. The non-inferiority.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-65 years)
* Infected with S. stercoralis (positive)
* Absence of major systemic illnesses
* Written informed consent

Exclusion Criteria:

* Any abnormal medical conditions or chronic disease
* Negative diagnostic result for S. stercoralis
* No written informed consent by the individual.
* Pregnant and lactating women.
* Recent use of an anthelmintic drug (within past 4 weeks)
* Attending other clinical trials during the study
* Known allergy to study medications (i.e. moxidectin, ivermectin)
* Currently taking medications with known interaction (i.e. for warfarin)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2022-02-05 (Actual); Primary Completion 2022-07-17 (Actual); Study Completion 2022-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Keiser, Prof. Dr, Principal Investigator — STPH
Locations (1):
- National Centre for Parasitology, Entomology and Malaria Control, Phnom Penh, Cambodia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sprecher VP, Hofmann D, Savathdy V, Xayavong P, Norkhankhame C, Huy R, Khieu V, Sayasone S, Hattendorf J, Keiser J. Efficacy and safety of moxidectin compared with ivermectin against Strongyloides stercoralis infection in adults in Laos and Cambodia: a randomised, double-blind, non-inferiority, phase 2b/3 trial. Lancet Infect Dis. 2024 Feb;24(2):196-205. doi: 10.1016/S1473-3099(23)00507-8. Epub 2023 Nov 7. PMID 37949090

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Moxidectin | Ivermectin
Started | 166 | 166
Completed | 154 | 161
Not Completed | 12 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moxidectin | Ivermectin | Total
Number analyzed (Participants) | 166 | 166 | 332
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (12.8) | 45.0 (12.7) | 44.9 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 86 | 165
  Male | 87 | 80 | 167
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Cambodia | 166 | 166 | 332
Strongyloides stercoralis infection intensity [Count of Participants; unit: Participants]
  Light | 102 | 103 | 205
  Moderate | 44 | 44 | 88
  Heavy | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Cure Rate Against Strongyloides Stercoralis
Description: The conversion from being larvae positive pre-treatment to larvae negative post-treatment, or cure rate (CR).
Time Frame: 14-21 days after treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Moxidectin | Ivermectin
Number analyzed (Participants) | 154 | 161
percentage of participants | 94.8 [90.0 to 97.7] | 99.4 [96.6 to 100]

2. Secondary Outcome: Larvae Reduction Rate (LRR) Against Strongyloidiasis Stercoralis
Description: Larvae per gram (LPG) stool sample will be assessed by calculating the mean of the larvae counts from the three duplicate Baermann assays and divided by the mean weighted amount of these stool samples. The LRR will be calculated following: (LRR = (1-(mean at follow-up/mean at baseline))*100)
Time Frame: 14-21 days after treatment. The originally planned follow-ups at 42-49 days and 63-70 days as well as the sample collection every second day between day 0 and day 70 (Moxidectin arm, n=50) was not performed.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | Moxidectin | Ivermectin
Number analyzed (Participants) | 154 | 161
percent change | 98.8 [96.0 to 99.9] | 100 [100 to 100]

3. Secondary Outcome: CRs Against Concomitant Soil-transmitted Helminth Infections - Ascaris Lumbricoides
Description: CRs will be calculated for Ascaris lumbricoides, Trichuris trichiura and hookworm infections as described in primary outcome.
Time Frame: 14-21 days after treatment
Population: No participants infected with Ascaris lumbricoides pre- or post-treatment
Arm/Group | Moxidectin | Ivermectin
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: CRs Against Concomitant Soil-transmitted Helminth Infections - Trichuris Trichiura
Description: as for outcome 3
Time Frame: 14-21 days after treatment
Population: No participants infected with Trichuris trichiura pre- or post-treatment
Arm/Group | Moxidectin | Ivermectin
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: CRs Against Concomitant Soil-transmitted Helminth Infections - Hookworm
Description: as for outcome 3
Time Frame: 14-21 days after treatment
Population: Participants co-infected with Hookworm
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Moxidectin | Ivermectin
Number analyzed (Participants) | 111 | 100
percentage of participants | 82.0 [74.7 to 89.2] | 81.0 [73.2 to 88.8]

6. Secondary Outcome: Number of Participants Reporting Adverse Events
Description: Participants will be monitored on site for at least 3 hours following treatment for any acute adverse events. In addition, participants will be interviewed 2-3 and 24 hours and at several weeks after treatment about the occurrence of adverse events. A standardized symptom questionnaire is used, that includes the recording of headache, abdominal pain, itching, nausea, vomiting, diarrhea, allergic reaction as well as any further mentioned event by the participant.
Time Frame: 2-3 hours, 24 hours and 14-21 days after treatment. The originally planned follow-ups at 42-49 days and 63-70 days after treatment were not conducted.
Population: Analysis population at 2-3 hours after drug administration: N=332. Analysis population at 24 hours after drug administration: N=332. Analysis population at 14-21 days after drug administration: N=315.
Measure: Count of Participants; unit: Participants
Arm/Group | Moxidectin | Ivermectin
Number analyzed (Participants) | 166 | 166
Participants
  2-3 hours: Headache | 4 | 10
  2-3 hours: Abdominal pain | 2 | 4
  2-3 hours: Itching | 3 | 0
  2-3 hours: Nausea | 0 | 0
  2-3 hours: Vomiting | 0 | 0
  2-3 hours: Diarrhea | 1 | 1
  2-3 hours: Allergic reaction | 0 | 0
  24 hours: Headache | 4 | 2
  24 hours: Abdominal pain | 1 | 1
  24 hours: Itching | 2 | 5
  24 hours: Nausea | 0 | 0
  24 hours: Vomiting | 0 | 1
  24 hours: Diarrhea | 0 | 1
  24 hours: Allergic reaction | 0 | 0
  14-21 days: Headache: number analyzed (Participants) | 154 | 161
  14-21 days: Headache | 0 | 0
  14-21 days: Abdominal pain: number analyzed (Participants) | 154 | 161
  14-21 days: Abdominal pain | 0 | 0
  14-21 days: Itching: number analyzed (Participants) | 154 | 161
  14-21 days: Itching | 0 | 0
  14-21 days: Nausea: number analyzed (Participants) | 154 | 161
  14-21 days: Nausea | 0 | 0
  14-21 days: Vomiting: number analyzed (Participants) | 154 | 161
  14-21 days: Vomiting | 0 | 0
  14-21 days: Diarrhea: number analyzed (Participants) | 154 | 161
  14-21 days: Diarrhea | 0 | 0
  14-21 days: Allergic reaction: number analyzed (Participants) | 154 | 161
  14-21 days: Allergic reaction | 0 | 0

7. Other Pre Specified Outcome: Socioeconomic Characteristics (SES)
Description: To all participating households, a brief questionnaire will be administered assessing information on socioeconomic characteristics (SES) and access to sanitation, water facilities, and hygiene behaviour.
Time Frame: Pre-treatment
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Genetic Profiling of S. Stercoralis Positive Stool Samples
Description: From all S. stercoralis positive stool samples, the extracted larvae will be stored in 70% Ethanol after examination by Baermann. Samples will be shipped to the investigating laboratory (La Trobe University) at room temperature.
Time Frame: Pre-treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 14-21 days
Description: Participants were monitored at the site for 3 hours following treatment. In addition, participants were interviewed at 2-3 and 24 hours after treatment and retrospectively at 14-21 days about the occurrence of adverse events.
  Since no adverse events were reported at 14-21 days post-treatment, the adverse events table contains the summary of events reported within 24 hours after drug administration.
Arm/Group | Moxidectin | Ivermectin
All-Cause Mortality (participants affected / at risk) | 0/166 | 0/166
Serious Adverse Events (participants affected / at risk) | 0/166 | 0/166
Other Adverse Events (participants affected / at risk) | 15/166 | 19/166
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moxidectin (N=166) | Ivermectin (N=166)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Allergic reaction (General disorders) | 0 (0) | 0 (0)
Headache (General disorders) | 8 (8) | 10 (12)
Nausea (General disorders) | 0 (0) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 4 (5) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-10): https://cdn.clinicaltrials.gov/large-docs/88/NCT04848688/Prot_SAP_000.pdf